CLINICAL TRIAL: NCT06241755
Title: Phase III Multi-center Randomized, Double-blind and Positive-controlled Clinical Trial for Evaluating the Efficacy and Safety of BCG for Therapeutic Use in the Prevention of Postoperative Recurrence of Medium/High-risk Non-muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Clinical Trial for Evaluating the Efficacy and Safety of BCG for Therapeutic Use in the Prevention of Postoperative Recurrence of Medium/High-risk Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu CoenBiotech Co., Ltd (Industry)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KN-BCG-III
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Non-Muscle Invasive Bladder Cancer
Keywords: Non-Muscle Invasive Bladder Cancer; Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — Therapeutic Uses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium-risk non-muscle invasive bladder cancer (NMIBC) (Experimental): Induction phase: Once weekly instillation for six consecutive times; Maintenance phase: Once every two weeks (Q2W) for three consecutive times and then once every four weeks (Q4W) for a total of 19 times.
  Interventions: Drug: BCG for Therapeutic Use
- High-risk non-muscle invasive bladder cancer (NMIBC) (Experimental): Induction phase: Once weekly instillation for six consecutive times; Maintenance phase: Once every two weeks (Q2W) for three consecutive times and then once every four weeks (Q4W) for a total of 19 times.
  Interventions: Drug: BCG for Therapeutic Use

INTERVENTIONS:
Drug: BCG for Therapeutic Use — Specification: 60 mg (6.0×10^7 CFU)/vial, each vial contains BCG 60 mg and each mg BCG shall have a count of live bacteria not less than 1.0×10^6 CFU.
  Usage & dosage: Dissolving two vials (120 mg) into 40-50 mL normal saline and shaking thoroughly. Following the procedures of surgical cauterization, inserting a Foley tube into cystic cavity and instilling diluted drug solution. After instillation, constantly changing body positions of a patient, such as left/right recumbent and supine/prostrate. Each position is maintained for around 30 min. Self-discharging drug solution after 2h.
  Other Names: BCG
Drug: BCG for Therapeutic Use — Specification: 60 mg/vial with a count of live BCG bacteria not less than 1.0×10^6 CFU/mg.
  Usage & dosage: Dissolving two vials (120 mg) into 40-50 mL normal saline and shaking thoroughly. Following the procedures of surgical cauterization, inserting a Foley tube into cystic cavity and instilling diluted drug solution. After instillation, constantly changing body positions of a patient, such as left/right recumbent and supine/prostrate. Each position is maintained for around 30 min. Self-discharging drug solution after 2h.
  Other Names: BCG

SUMMARY:
A phase III multi-center randomized, double-blind and positive-controlled clinical trial for evaluating the efficacy and safety of BCG for Therapeutic Use（BCG） in the prevention of postoperative recurrence of medium/high-risk non-muscle invasive bladder cancer (NMIBC).

DETAILED DESCRIPTION:
Instillation of BCG for Therapeutic Use（BCG） into the urinary bladder (intravesical administration) improves rates of tumor recurrence and progression after adequate transurethral resection of bladder (TURBt) of moderate to high risk, non-muscle-invasive bladder cancer (NMIBC).

To determine the efficacy and safety of BCG as an adjuvant therapy method in patients with NMIBC., we conduct a randomized, double-blinded, positive controlled phase 3 clinical trial. The target population is adults with moderate to high risk NMIBC (Ta ，T1 or tis) suitable for intravesical BCG treatment. Key eligibility criteria include prior transurethral resection of all visible tumor, adequate organ function, and ECOG performance status 0-2. 412 Subjects will be administrated with 120mg Intravesical BCG. The treatment includes Induction perfusion period (weekly x 6), followed by maintenance perfusion period (Q2W x 3 times ,then once monthly). totaled with 19 times BCG perfusion, and lasting until 1 year after surgery. The primary endpoint is 1-year recurrence-free survival rate.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients aged ≥18 year and ≤75 year
* 2. According to the stipulations of Guidelines on Diagnosing & Treating Bladder Cancer (Edition 2022) as promulgated by National Health Commission, an initial definite diagnosis of medium/high-risk non-muscle invasive urothelial bladder cancer (T1/Ta/Tis) as confirmed by histological examination and requiring an adjuvant therapy of BCG bladder instillation；
* 3. After a thorough TURBt, all tumors should be grossly invisible. Patients requiring a second procedure are also eligible for inclusion. Those fulfilling the requirements of a second procedure may do so. Patients fulfilling the requirements of a second procedure shall meet the following criteria:

  1. Criteria of a second TURBt: 1) Initial TURBt is insufficient; 2) No muscular specimen during an initial TURBt; 3) Stage T1 tumor; 4) G3 (advanced grade) tumor, except for simple in situ tumor;
  2. A second TURBt is recommended within Weeks 2-6 after an initial procedure. It is optimal at Week 4. After TURBt until BCG bladder instillation, no other instillations are allowed except for 1st/2nd immediate instillation chemotherapeutic agents. For the last TURBt, only epirubicin is reserved for immediate instillation chemotherapy;
  3. Subjects undergoing a second TURBt and starting BCG therapy at Weeks 2-4 after a second procedure;
  4. Based upon the first/second result of histopathology examination, comprehensively evaluating whether or not a certain patient is eligible for inclusion.
* 4. A previous history of never receiving any therapy of BCG bladder instillation;
* 5. ECOG score: 0-2 points;
* 6. Clinical laboratory tests fulfilling the following features:

  1. Blood routine: Within Day 14 prior to randomization, never using any hematopoietic growth factor or blood transfusion, including absolute neutrophil count (ANC) ≥1500/mm3 or ≥1.5×109/L; platelet ≥100000/mm3 or 100×109/L; hemoglobin ≥9 g/dL.
  2. Liver function: total serum bilirubin ≤1.5× upper limit of normal (ULN); for subjects with Gilbert syndrome total serum bilirubin <3×ULN ;AST/ALT ≤2.5×ULN.
  3. Renal function: defined as estimated creatinine clearance ≥50 mL/min according to the formula of Cockcroft-Gault;
  4. Blood coagulation function: APTT ≤ 1.5×ULN and INR ≤1.5×ULN.
* 7. Capable of understanding the procedures and methods of clinical study and participating voluntarily after offering thorough informed consents.

Exclusion Criteria:

* 1. Current users of immune suppressants, hormones or radiotherapy and potentially causing systemic BCG-related disease responses (patients requiring an injection of matching hormones after thyroidectomy or adrenalectomy are also eligible for inclusion);
* 2. Allergic to BCG or its analogues;
* 3. Presence of active TB lesions, currently receiving an anti-TB therapy or taking any anti-TB regimen within Month 6 prior to screening;
* 4. Known or suspected intraoperative bladder perforation;
* 5. Presence of severe gross hematuria pre-dosing as judged by investigators and with a suspicion of non-healing surgical wound;
* 6. Presence of concurrent cystitis with such signs of cystic irritation as urinary frequency/urgency/pain as judged by investigators or previously receiving therapies of other bladder instillation drugs and irritating bladder signs severe enough to interfere with study evaluations;
* 7. Individuals with a previous history of such severe adverse events as BCG sepsis or systemic infections;
* 8. Complete cystic urinary incontinence is defined as using six and more pads with 24h;
* 9. Concurrently with other urogenital system tumors or other malignant solid organ tumors;
* 10. Individuals with a previous history of severe cerebrocardiovascular, pulmonary, hepatic and renal diseases or hypertension and diabetes mellitus clinically uncontrollable as judged by investigators;
* 11. Individuals with an evidence of focal advanced or metastatic muscular infiltration urothelial cancer or concurrent extra-cystic non-muscle invasive urothelial transition cell cancer;
* 12. Receiving chemotherapy, radiotherapy or immunotherapy within Week 4 prior to an initial dose (except for immediate postoperative intravesical chemotherapy);
* 13. Pregnant or lactating women;
* 14. Individuals failing to adopt effective birth control measures during study until Month 6 after the last dose;
* 15. Participating in a clinical study of another drug within Month 3 prior to screening;
* 16. Known dependents of opioids or alcohol;
* 17. Any of the following items: Positive antibodies of (HIV, treponema pallidum and acute/chronic active hepatitis B (HBsAg); copy number of HBV-DNA in peripheral blood ≥103/mL; HCV antibody positive with copy number of HCV ≥103 /mL;
* 18. Individuals with mental retardations or poor compliance;
* 19. Any circumstance potentially boosting subject risks or interfering with study implementations as judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence-free survival (1-year RFS%): | 1 year
  Evaluating the percentage of subjects staying free from recurrence or mortality from randomized to Year 1 (first occurring as a priority)

SECONDARY OUTCOMES:
2-year recurrence-free survival (2-year RFS%) | 2 year
1-year progression-free survival (1-year PFS%) | 1 year
2-year progression-free survival (2-year PFS%) | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No